CLINICAL TRIAL: NCT04172571
Title: An Open-Label Multi-Center Phase Ib/II Study of the Combination of AK105 and Anlotinib Hydrochloride in the First-Line Treatment of Patients With Unresectable Hepatocellular Carcinoma
Brief Title: A Study of the Combination of Anti-PD-1 AK105 and Anlotinib in First-line Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akeso Tiancheng, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK105-203
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: VEGF; Anti-PD-1; Tyrosine Kinase Inhibitor (TKI); Angiogenesis-related kinases
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AK105 and anlotinib (Experimental)
  Interventions: Biological: AK105; Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Biological: AK105 — Anti-PD-1 antibody; IV infusion, 200 mg Q3W
Drug: Anlotinib Hydrochloride — multi-targeted receptor TKI; oral administration; every 3 weeks as one cycle administered as 2 weeks on/1 week off

SUMMARY:
This is a multi-center,open-label study to evaluate the efficacy and safety of anti-PD-1 antibody AK105 plus anlotinib hydrochloride in the first-line treatment of patients with unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form voluntarily.
* Male or female，age over 18 years old (inclusive) and not more than 75 years old (inclusive), when signing the ICF.
* Expected life expectance ≥ 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
* Confirmation either by histology unresectable hepatocellular carcinoma..
* BCLC stage C, and non-resectable BCLC stage B .
* No prior systemic therapy for HCC.
* Child-Pugh class A and B (≤7 points).
* At least one measurable lesion according to RECIST criteria.
* Adequate hematologic and end-organ function.
* For women of childbearing potential: agreement to remain abstinent; For men: agreement to remain abstinent.

Exclusion Criteria:

* Prior treatment with anti-PD1, anti-PD-L1 or anti-CTLA-4 antibody therapy.
* Active ongoing infection requiring therapy.
* History of severe hypersensitivity reaction to another monoclonal antibody.
* Received any live attenuated vaccine within the last 30 days.
* Other malignancy requiring treatment in the prior 5 years with the exception of locally treated squamous or basal cell carcinoma.
* Pregnant, breast feeding, or planning to become pregnant.
* Active or prior documented autoimmune or inflammatory disease with some exceptions.
* Central nervous system metastases and/or carcinomatous meningitis.
* Medical condition that requires chronic systemic steroid therapy, or any other form of immunosuppressive medication.
* Co-infection of HBV and HCV.
* Inadequately controlled arterial hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to approximately 18 months
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1.

SECONDARY OUTCOMES:
Number of subjects experiencing adverse events (AEs) | From the time of informed consent through 90 days after last dose of AK105
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Duration of response (DoR) | up to approximately 18 months
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Disease control rate (DCR) | up to approximately 18 months
  DCR is defined as the proportion of subjects with CR, PR, or SD based on RECIST v1.1.
Progression-free survival (PFS) | up to approximately 18 months
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Overall survival (OS) | up to approximately 24 months
  OS is the time from the date of first dosing to death due to any cause.
Observed concentrations of AK105 | From first dose of AK105 through 90 days after last dose of AK105
  The endpoints for assessment of PK of AK105 include serum concentrations of AK105 at different timepoints after AK105 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK105 through 90 days after last dose of AK105
  The immunogenicity of AK105 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Shunchang Jiao, MD, Principal Investigator — Chinese PLA General Hospital; Li Bai, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Pang X, Zhong T, Qu T, Chen N, Ma S, He X, Xia D, Wang M, Xia M, Li B. Penpulimab, an Fc-Engineered IgG1 Anti-PD-1 Antibody, With Improved Efficacy and Low Incidence of Immune-Related Adverse Events. Front Immunol. 2022 Jun 27;13:924542. doi: 10.3389/fimmu.2022.924542. eCollection 2022. PMID 35833116
- [Derived] Han C, Ye S, Hu C, Shen L, Qin Q, Bai Y, Yang S, Bai C, Zang A, Jiao S, Bai L. Clinical Activity and Safety of Penpulimab (Anti-PD-1) With Anlotinib as First-Line Therapy for Unresectable Hepatocellular Carcinoma: An Open-Label, Multicenter, Phase Ib/II Trial (AK105-203). Front Oncol. 2021 Jul 13;11:684867. doi: 10.3389/fonc.2021.684867. eCollection 2021. PMID 34327136